CLINICAL TRIAL: NCT06280066
Title: An Intervention-based Approach to Strengthen Life Skills and Psychological Resilience of Children With Cystic Fibrosis and Their Mothers
Brief Title: An Intervention-Based Approach to Strengthen the Psychological Health of Children With Cystic Fibrosis and Their Mothers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Selin Soyunmez, Research Assistant, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/607
Record Dates: First submitted 2024-01-05; First posted 2024-02-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis; Children; Resilience,Psychological; Laughter Yoga; Laughter Therapy; Mothers; Psychological Health; Lung Functions
Keywords: cystic fibrosis; children; psychological resilience; laughter yoga; laughter therapy; mothers; psychological health; lung functions
MeSH Terms: conditions — Cystic Fibrosis; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Children Intervention Group (Experimental): Intervention Program Based on Strengthening Psychological Resilience for Children with Cystic Fibrosis and Their Mothers. The program will be implemented for 10 weeks, with a total of 10 sessions, 1 session per week (each session consists of 2 sessions).
  Interventions: Other: Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers
- Mothers Intervention Group (Experimental): Intervention Program Based on Strengthening Psychological Resilience for Children with Cystic Fibrosis and Their Mothers. The program will be implemented for 10 weeks, with a total of 10 sessions, 1 session per week (each session consists of 2 sessions).
  Interventions: Other: Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers
- Children Controlled Group (No Intervention): No intervention.
- Mothers Controlled Group (No Intervention): No intervention.

INTERVENTIONS:
Other: Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers — The content of the Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers will include the Psychological Resiliency Program for Children and Adolescents developed by Akar (2018), laughter yoga, meditation, breathing exercises and therapeutic story sessions.
  Arms: Children Intervention Group; Mothers Intervention Group

SUMMARY:
Cystic fibrosis (CF) is a life-threatening exocrine gland disease that is often diagnosed in childhood, and its incidence tends to increase and affect physical and mental health.The purpose of this study is to evaluate the effectiveness of the Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers, prepared for children with CF (8-12 years old) and their mothers.In the first stage, the CF experiences of children with cystic fibrosis and how they perceive these experiences will be examined with visual phenomenology, and their mothers' CF experiences and perceptions will be examined with phenomenology. In this regard, 10 children will be asked to draw pictures and their pictures will be analyzed. In-depth individual interviews will be held with mothers.In the 2nd stage, the effectiveness of the Intervention Program Based on Strengthening Psychological Resilience for Children Diagnosed with Cystic Fibrosis and Their Mothers will be determined with a pre-test-post-test randomized controlled experimental design.In the literature review, Gpower analysis was performed (α: 0.05, β: 0.99, d: 1.88) based on the results of studies conducted with children diagnosed with CF and their parents, similar to this study, and 15 samples were used for each group. It is planned to recruit people. Considering the possibility of data loss in the study, it was always deemed appropriate to include 22 people for the group. It was planned to sample a total of 88 children with CF and their mothers, 44 in the intervention group and 44 in the control group. In the 3rd stage, after the experiment, the participants' experiences regarding the intervention program will be examined through interviews and qualitative research method. Thus, qualitative interviews will be conducted before and after the experiment. Data will be collected using these tools: Children; Child and Mother Descriptive Characteristics Form, Semi-Structured Interview Form,Respiratory Function Test, Reorganized Cystic Fibrosis Questionnaire, Psychological Resilience Attitude and Skills Scale and Functional Disability Inventory; Mothers; The Revised Cystic Fibrosis Questionnaire, The Depression Anxiety and Stress Scale, Post-Traumatic Growth Scale and Brief Psychological Resilience Scale. Measurements will be taken before the intervention, after the intervention, at the 1st and 3rd months.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a life-threatening exocrine gland disease that is often diagnosed in childhood and its incidence tends to increase. CF affects many systems, especially the respiratory and gastrointestinal systems, and is life-threatening with its progressive course. In addition to the complications that arise due to the disease affecting many systems, the limited life expectancy and poor prognosis also bring psychological and social problems for children and their families. Especially if it is a genetically inherited disease, it may cause the parent to blame himself or herself and experience psychological problems. It is stated that in order to make it easier for children with CF and their families to cope with the negativities brought about by the disease, their psychological resilience levels should be strengthened and health professionals should encourage families to do so. Apart from increasing the level of psychological resilience, other methods that contribute to the reduction of psychological problems include yoga, meditation and laughter yoga. Laughter yoga is a series of exercises that combine gratuitous laughter with yoga breathing techniques, as well as stretching-relaxation techniques, laughter and deep breathing exercises. It is reported that laughter yoga physiologically increases breathing in the body, relaxes muscles, strengthens mental function by reducing the level of stress hormones, reduces burnout, depression and anxiety levels, positively affects the quality of life and increases psychological well-being. In this context, an intervention program was created for children with CF and their mothers, including psychological resilience training, laughter yoga, concentrated breathing exercise and meditation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Children:

* Being between the ages of 8-12,
* FEV 1 value, which is considered as the acceptance criterion in the terminal period in cystic fibrosis, is over 40%,
* Not having any physical or mental disability,
* Ability to communicate in Turkish,
* Not having an additional diagnosis such as type 1 diabetes or phenyl ketonuria,
* Volunteering to participate in the research.

Inclusion Criteria for Mothers:

* Having a child diagnosed with CF between the ages of 8-12,
* Not having any physical or mental disability,
* Ability to communicate in Turkish,
* Volunteering to participate in the research.

Exclusion Criteria:

Exclusion Criteria for Children:

* Being on mechanical ventilation,
* Being in the preparation phase for lung transplantation
* Failure to fully participate in the Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers.

Exclusion Criteria for Mothers:

* Lack of internet connection at home,
* Failure to fully participate in the Intervention Program Based on Strengthening the Psychological Resilience of Children Diagnosed with Cystic Fibrosis and Their Mothers.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The Respiratory Function Test | The measurement will start two weeks before the intervention, immediately after the intervention.
  Children will have a respiratory function test performed at the center where the research will be conducted. As a result of the rest, the children's FEV1 and FVC values will be examined.
The Revised Cystic Fibrosis Questionnaire Child Form | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  The scale that evaluates the quality of life due to the impact of cystic fibrosis-specific health status is a 4-point Likert type. A higher score indicates a better CF-specific health-related quality of life.
Psychological Resilience Attitude and Skills Scale Child Form | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  Scores range from 34 to 136 on the scale, and as the score increases, the level of psychological resilience of children increases.
Functional Disability Inventory Child | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  It is a child self-report tool that evaluates the impact of the disease on physical and psychosocial functioning in daily social roles and daily activities at home and at school. The scale is a 5-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 60. As the score obtained from the scale increases, the level of disability increases.
The Revised Cystic Fibrosis Questionnaire Parent Form | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  The CFQ-R Parent version is a self-report instrument consisting of 44 items grouped into 11 domains assessing physical functioning, emotional functioning, vitality, school performance, eating disorders, weight, body image, treatment burden, health perceptions, and respiratory and digestive symptoms. A higher score on the CFQ-R Parent version indicates a better CF-specific health-related quality of life.The total point range is 0-100, with higher scores indicating better CF-specific health-related quality of life.
Depression Anxiety and Stress Scale | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  It will be used to determine mothers' depression, anxiety, and stress levels. The scale is a 4-point Likert type and consists of 3 subscales (depression, anxiety, and stress) and 21 questions. The minimum score that can be obtained from the scale is 0, and the maximum score is 21. A high score on the sub-dimension of the scale indicates that the level of that sub-dimension is high.
Post-Traumatic Growth Scale | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  As the score obtained from this scale, which will be used to determine the post-traumatic growth levels of mothers, increases, the post-traumatic growth level also increases.The scale is a 6-point Likert-type scale, consisting of 5 sub-dimensions and a total of 21 items. The minimum score that can be obtained from the scale is 0, and the maximum score is 105. As the score increases, the level of post-traumatic growth also increases.
Brief Psychological Resilience Scale | The measurement will start two weeks before the intervention, immediately after the intervention, and 1 and 3 months after the intervention.
  A minimum of 6 and a maximum of 30 points can be obtained from this scale, which will be used to determine the psychological resilience levels of mothers, and higher scores indicate higher psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Sezer Efe, Principal Investigator — TC Erciyes University; Selin Söyünmez, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No